CLINICAL TRIAL: NCT07104864
Title: High Efficiency of Early Detection of Synchronous Pancreatic Ductal Adenocarcinoma in Patients With Chronic Pancreatitis
Brief Title: Early Detection of PDAC in Patients With Chronic Pancreatitis
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: ZXIITYFY2024202
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Chronic Pancreatitis; PDAC - Pancreatic Ductal Adenocarcinoma
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: histopathological confirmation — histopathological confirmation

SUMMARY:
The goal of this study is to find simple warning signs that doctors can use to spot pancreatic cancer early in people who have chronic pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

1. a confirmed diagnosis of chronic pancreatitis; (2) availability of pathological confirmation.

Exclusion Criteria:

1. age less than 18 years; (2) ambiguous pathology, including cases with only cytological findings or indications of pancreatic tissue alone; (3) preoperative diagnosis of PDAC or other pancreatic tumors before invasive procedure; (4) presence of tumors in other organs; (5) patients with missing data exceeding 15% of the total dataset.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with CP upon admission to the First Affiliated Hospital of Xi'an Jiaotong University between January 2013 and December 2023
Sampling Method: Non-Probability Sample
Enrollment: 359 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
pathological diagnosis of PDAC | January 2013 and December 2023

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided